CLINICAL TRIAL: NCT02488096
Title: Improving Prostate Cancer Detection Using MRI-Targeted TRUS-Guided Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REB15-27
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRUS-Guided Biopsy (Active Comparator): Transrectal Ultrasound (TRUS)-guided biopsy systematic 12-core biopsy (standard care)
  Interventions: Device: TRUS-Guided Biopsy
- MRI + TRUS-Guided biopsy (Experimental): Prostate MRI later followed by systematic 12-score TRUS-guided biopsy + targeted biopsy of additional MRI-detected scores.
  Interventions: Device: MRI + TRUS-Guided Biopsy

INTERVENTIONS:
Device: TRUS-Guided Biopsy — The standard care TRUS-guided biopsy is a schematic 12 core biopsy scheme with 2 cores taken from each of standard 6 zones. In some cases, the radiologist may take additional cores beyond 12 if suspicious areas are suspected from clinical findings or TRUS. TRUS-guided biopsies will be performed by a designated group of radiologists. An overall score out of 5 of likelihood of clinically significant prostate cancer will be recorded for each individual patient. The biopsy will be scheduled within 1 week of referral.
  Other Names: Transrectal Ultrasound Guided Biopsy
  Arms: TRUS-Guided Biopsy
Device: MRI + TRUS-Guided Biopsy — A designated radiologist will perform all MRI exams. The radiologist will identify locations of the prostate gland of the standard 12 cores to be taken and any additional lesions deemed to be suspicious for cancer.
  The procedure for the MRI-targeted biopsy will be exactly the same as the TRUS-guided biopsy except that an additional 2 cores per area may be taken beyond the standard 12 cores in areas that were previously identified by MRI on the map. The systematic 12-core biopsy will always be performed first. The radiologist performing the MRI-targeted biopsy will review the MRI targets prior to the biopsy as per standard of care, and he/she will also perform the TRUS-guided biopsies for this group. Patients will be scheduled for their biopsy ~ 1 week after the MRI.
  Other Names: Magnetic Resonance Imaging + MRI-Targeted TRUS-guided Biopsy
  Arms: MRI + TRUS-Guided biopsy

SUMMARY:
The purpose of this study is to determine if using MRI can improve cancer detection by identifying potential cancer targets prior to TRUS-guided biopsy in populations that have previous inconclusive results from TRUS-guided biopsies.

DETAILED DESCRIPTION:
Accurately diagnosing clinically significant prostate cancer at a time when the benefits of treatment outweigh the harm continues to elude clinicians because of the complex nature of prostate cancer. When patients are found to have a high prostate specific antigen (PSA) blood test, an abnormal digital rectal exam, or they have prostate cancer but are delaying treatment (active surveillance), they are referred for transrectal ultrasound (TRUS) guided biopsy. The sensitivity of TRUS with 12-core biopsies is only 53-68% so cancers can be missed, particularly in the anterior region of the prostate. In some cases, TRUS can be used to rule out other causes of abnormal test findings, however the specificity of TRUS is also fairly poor making it difficult for a man to know for certain if he is cancer free. Unfortunately, biopsies also cause serious side effects including incontinence, bowel dysfunction, infection and pain. Increasing the number of cores taken during biopsy does not typically translate to better detection rates.

Magnetic resonance imaging (MRI) has much greater resolution than TRUS and can therefore, detect changes in the prostate more accurately. If conducted prior to a targeted biopsy, MRI can also reduce the number of cores taken compared to a standard biopsy (e.g. 2-4 cores vs. 12 cores), which could reduce biopsy side effects while simultaneously increasing detection of clinically significant cancer compared to routine 12-core biopsies and saving health care system dollars. Technology that combines MRI at the same time as biopsy (MRI-TRUS fusion biopsy) is increasingly being used, with some promising results. However, these techniques require expensive equipment and specially-trained personnel, and are more time-consuming and restrictive in when the procedure can occur. Utilizing MRI prior to a TRUS-guided biopsy could provide the same benefits in terms of cancer detection, but at a more reasonable cost and shorter wait-times as MRI alone can be done in a variety of settings and times.

If the results of this study demonstrate that MRI-targeted biopsy improves detection of clinically significant cancer over TRUS-guided biopsy alone, it would suggest that this protocol may be a more practical solution. Moreover, if the results show that MRI-targeted biopsy could reduce the number of cores taken without missing clinically significant cancers, the local biopsy protocol could be adjusted in the future to minimize unnecessary harm in these populations of men. In summary, this study will have practical merits in minimizing costs and patient morbidity associated with unnecessary prostate biopsies and treatments across Canada.

The primary objective of this study is to determine if using MRI can improve cancer detection by identifying potential cancer targets prior to TRUS-guided biopsy in populations that have previous inconclusive results from TRUS-guided biopsies.

The secondary objectives are to:

* Determine the sensitivity, specificity, positive and negative predictive value of MRI in predicting clinically significant prostate cancer
* Identify areas of the prostate that would benefit most from MRI
* Estimate Type 1 and Type II errors of using MRI-targeted biopsy samples compared to both MRI-targeted and standard 12-core.
* Estimate cost savings by using MRI-targeted biopsy samples only compared to both MRI-targeted and standard 12-core.
* Compare cost-effectiveness of using MRI prior to TRUS-guided biopsy compared to MRI-fusion biopsy used in other centers

This is a prospective, single institution randomized clinical controlled trial.. Participants will be randomized in a 1:1 ratio to one of the following groups:

1. Control Group: TRUS-guided systematic 12-core biopsy (standard care)
2. Experimental Group: prostate MRI later followed by systematic 12-core TRUS-guided biopsy + targeted biopsy of additional MRI-detected cores

ELIGIBILITY:
Inclusion Criteria:

* Referred for an ultrasound-guided prostate biopsy
* Indication 1: Men without a history of prostate cancer referred to the PAC for a biopsy who have a history of 1 negative biopsy who are being referred for a follow-up biopsy
* Indication 2: Men who have a history of diagnosis of prostate cancer and are currently on active surveillance under the care of an oncologist who are referred to the PAC for a follow-up biopsy

Exclusion Criteria:

* Are unable to consent on their own behalf
* Less than 3 months since previous biopsy (to avoid inflammation and hemorrhage confounding MRI image)
* A history of treatment for prostate cancer (including surgery, chemotherapy or radiotherapy)
* Emergent/urgent biopsy referrals
* History of urinary tract infections or prostatitis in the last 3 months
* Contraindications to MRI:
* Ferromagnetic or otherwise non-MRI compatible aneurysm clips
* The presence of an implanted pacemaker or implanted defibrillator device
* Contraindication to receiving Gadolinium containing contrast for the which may include past or current kidney disease or injury or kidney transplant
* Severe claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Clinically Significant Cancer Detection (Biopsy) | participants will be followed until diagnosis, an expected average of 2 weeks
  * max core length >=3mm (Epstein criteria)
  * Gleason score >=3+4 (Epstein criteria)
  * clinical Stage T2c (D'Amico criteria)
  * Gleason score 6 with >50% involvement of prostate

SECONDARY OUTCOMES:
Clinically Significant Cancer Detection (Prostatectomy) | Up to 6 months after enrollment
  Clinically significant cancer detected at prostatectomy using the same criteria as the primary outcome. Prostatectomy can reveal slightly different outcomes than biopsy so these data will be gathered to determine the true positive and negative predictive value of the MRI using whole-mount specimens.
Proportion of Men Who Could Have Potentially Avoided Biopsy | participants will be followed until diagnosis, an expected average of 2 weeks
  * Determined by specificity and negative predictive values.
  * Negative predictive value will be defined as the ratio of patients with a MRI suspicion score ≤2 to patients with clinically insignificant disease.
Proportion of Cancers Correctly Identified by MRI | participants will be followed until diagnosis, an expected average of 2 weeks
  - An MRI cancer risk score of ≥4 for each core will be used to designate a positive test for predicting positive cancer in each core and ≤2 to designate a negative test for predicting no cancer.
Proportion of Cancers that would have been Missed | participants will be followed until diagnosis, an expected average of 2 weeks
  Proportion of cancers that would be have been missed if only cores from targeted biopsy had been taken instead of systematic 12-core biopsy
Estimated difference in cost | participants will be followed until diagnosis, an expected average of 2 weeks
  Estimated difference in cost by using MRI-targets only in biopsy vs systematic 12-core

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer St. Onge, PhD, Principal Investigator — Research, Regina Qu'Appelle Health Region; Ashok Verma, MB, Principal Investigator — Radiology, Regina Qu'Applle Health Region
Locations (1):
- Regina Qu'Appelle Health Region, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No